CLINICAL TRIAL: NCT03070366
Title: Randomized Phase II Trial Comparing Chemotherapy Combined With Stereotactic Radiotherapy and Stereotactic Radiotherapy Alone, for Treatment of Oligometastases in Squamous Cell Cancers of the Upper Aerodigestive Tract
Brief Title: Stereotactic Radiotherapy Combined With Chemotherapy or Not for Treatment of Oligometastases in HNSCC
Acronym: OMET
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Groupe Oncologie Radiotherapie Tete et Cou (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: GORTEC 2014-04
Record Dates: First submitted 2017-01-16; First posted 2017-03-03 (Actual); Last update posted 2025-09-02 (Actual); Status verified 2025-08

CONDITIONS: Head and Neck Squamous Cell Carcinoma
Keywords: Oligometastasis; stereotactic irradiation
MeSH Terms: conditions — Squamous Cell Carcinoma of Head and Neck | interventions — Drug Therapy; Radiosurgery

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Chemotherapy combined with stereotactic radiotherapy (RT) (Active Comparator): Chemotherapy is based on patient Performance Status (PS) and comorbidities:
  * PS 0-1: standard treatment: 6 cycles, every 3 weeks cisplatin (100 mg/m² iv on D1), 5FU (4000 mg/m² total dose starting on Day 1 to Day 4 and during 96h in continuous infusion)
  * PS 2/cardiac contra-indication to 5 Fluorouracil (5FU): 6 cycles, every 3-4 weeks cisplatin (100 mg/m² iv on Day 1) or carboplatin Area Under Curve (AUC) 4 or 5 on Day 1 In both case: Cetuximab (loading dose 400 mg/m² iv on Day1, then 250 mg/m² weekly or 500mg/m² every 2 weeks).
  Cycle 1 of systemic treatment will be administered before the start of the stereotactic RT. Then, following cycles will be performed after the end of stereotactic irradiation.
  Cetuximab maintenance: 250 mg/m² iv weekly. It will be given only if at least disease stabilization is observed at the end of chemotherapy, and will be continued until progression or unacceptable toxicity.
  Interventions: Drug: Chemotherapy; Radiation: Stereotactic radiotherapy
- stereotactic radiotherapy (Experimental): Splitting will be based on the tumor diameter, and proximity of organs at risk which constitutes any limiting toxicities. It will be 3 or 5 fractions based on the recommendations (CARO-Stereotactic Body Radiation Therapy (SBRT) 2012) and for the purpose of harmonization practices. The prescription dose is 3 x 10 = 30 Gy 3 x 11 = 33 Gy or 3 x 15 = 45 Gy (if 3 fractions) with the possibility of 3 x 20 Gy to the peripheral lung nodules with tracking in Cyberknife or 5 x 7 = 35 Gy or 5 Gy x 10 = 50 (if 5 fractions). Beyond 3 cm of tumor diameter and / or to a distance of less than 1 cm from the GTV in an organ critical risk (eg spinal cord), a splitting up into 5 sessions must be privileged.
  Interventions: Radiation: Stereotactic radiotherapy

INTERVENTIONS:
Drug: Chemotherapy — * cisplatin
  * 5FU
  * carboplatin
  * cetuximab
  Arms: Chemotherapy combined with stereotactic radiotherapy (RT)
Radiation: Stereotactic radiotherapy — Stereotactic radiotherapy

SUMMARY:
The aim of this study is to evaluate the rate of living patients at 1 year with a quality of life criteria (no decrease) and reduced toxicities. This criteria will be compared in both groups., A cost effectiveness study is scheduled also.

DETAILED DESCRIPTION:
Patients with cancers of aerodigestive tract have metastases limited in their evolution and a pauci-metastatic disease. In these cases, systemic therapy is the standard attitude. However, patients often received chemotherapy in their history and response rates are relatively low. The median survival is between 7 and 11 months with secondary effects and degradation of quality of life. It is a palliative treatment. Data on systemic treatment in the context of a micro-metastatic disease are limited. In contrast, stereotactic irradiation in pauci-metastatic context leads to better local control rates and may sustainedly reduce the progression of metastatic disease.

Stereotactic radiotherapy is increasing use in clinical practice for limited metastatic stages (oligo metastatic with 1-3 synchronized metastases). Radiotherapy in this indication has major advantages and a similar efficacy compared with other ablative treatments.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years
* PS:0-2
* Estimated life expectancy ≥ 6 months
* Histologically confirmed diagnosis of squamous cell carcinoma of the head and neck
* Target metastases can be treated in stereotactic radiotherapy
* 1-3 synchronized metastases with unrestricted anatomic site
* Greater cumulative diameter of synchronous metastases in once organ (liver, lung or brain) ≤ 6 cm with GTV = Clinical Target Volume (CTV)
* Global maximum diameter (GTV) allowed for pulmonary oligometastases (less than 2 cm from the mediastinum), brain, node, is ≤ 3cm
* Implementation of a method for taking into account movements and uncertainties (IGRT) for limiting the margin of CTV to PTV (PTV) so as not to exceed 7 cm large cumulative diameter of PTV
* Performing a positron emission tomography with 18F-2-fluoro-2-deoxy-D-glucose (FDG-PET) 4 weeks before the inclusion
* In case of cerebral metastases, MRI diagnostic is required
* If locoregional disease is treated, controlled and non-progressive for more than three months (+/- 4 weeks) at baseline, synchronized initial tumor is possible
* If metachronous metastases, locoregional disease previously treated should be monitored and considered not progressive for more than three months at baseline
* In case of prior cancer other than HNSCC, complete remission for over 5 years is possible, any biopsy of metastases is left to the appreciation of referring physician
* No chemotherapy or local treatment of metastases in the previous 6 months
* Laboratory tests consistent with the achievement of chemotherapy: Leukocytes> 3,000 / mm3 (including polynuclear> 2000 / mm3) platelets> 150,000 / mm3, serum glutamate oxaloacetate transminase (SGOT), serum glutamate pyruvate transaminase (SGPT), alkaline phosphatase, bilirubin <2.5 upper limit of normal (ULN)
* Affiliation to an health insurance
* Informed Consent Form signed

Exclusion Criteria:

* Concomitant participation in other interventional clinical trial within 4 weeks before inclusion
* Other prior ablative treatment of targets metastases (surgery, radio frequency) in the previous six months
* metachronous primitive tumor (second cancer) uncontrolled.
* contraindication to any systemic therapy (chemotherapy and / or targeted therapy)
* Known hypersensitivity reaction to 5FU, cisplatin, carboplatin, platin or cetuximab
* Active infection (infection requiring IV antibiotics), including active tuberculosis and known and declared human immunodeficiency virus (HIV)
* Other malignancies within 5 years prior to randomization, with the exception of adequately treated basal skin cancer and carcinoma in situ of the cervix
* Individual deprived of liberty by judicial or administrative decision, or under any kind of guardianship
* Pregnant or breast feeding women. Every woman who has childbearing potential, must have a negative pregnancy test (serum or urine) within 14 days previous treatment. Patients (men or women) must use a reliable method of contraception throughout treatment and for at least 6 months after discontinuation of chemotherapy.

Ages: 18 Years to 77 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 78 (Estimated)
Dates: Start 2015-09-21 (Actual); Primary Completion 2026-07 (Estimated); Study Completion 2026-07 (Estimated)

PRIMARY OUTCOMES:
Overall Survival without quality of life deterioration | 1 year
  Overall Survival rate without definitive deterioration of quality of life (by QLQC30) measured at 1 year post treatment

SECONDARY OUTCOMES:
Overall Survival | 1 year
Progression free survival | through study completion, an average of 1 year
Number of participants with adverse events grade 3 as assessed by CTCAE v4.0 within the first 6 months of treatment | up to 6 months
  Toxicity of grade > or equal to 3, occurring within the first 6 months of treatment
Number of participants with treatment related adverse events as assessed by CTCAE v4.0 | through study completion, an average of 1 year
Overall response rate | through study completion, an average of 1 year

CONTACTS AND LOCATIONS:
Locations (1):
- Hôpital Nord Franche Comté, Montbéliard, France

IPD SHARING:
Plan to Share IPD: Yes
The Data Monitoring Committee will meet every year either by a physical meeting or by conference call. Data on the recruitment, toxicity and autonomy are submitted every year.